CLINICAL TRIAL: NCT00612677
Title: Phase II Combination of Pemetrexed and Oxaliplatin in Patients With Recurrent Non-Small Cell Lung Cancer After Failure to Platinum Based Adjuvant Chemotherapy
Brief Title: Pemetrexed &Oxaliplatin in Patients w Recurrent NSCLCa After Failure to Platinum Based Adjuvant Chem
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual - the 1 patient accrued did not go on treatment
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15010; OX-04-006 (Other Grant/Funding Number: Sanofi-Aventis US, Inc.)
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Results first posted 2011-04-20 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2013-12

CONDITIONS: Lung Cancer
Keywords: recurrent; non-small cell
MeSH Terms: conditions — Lung Neoplasms; Recurrence | interventions — Oxaliplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Premetrexed and Oxaliplatin (Experimental): Patients will be treated with oxaliplatin 120 mg/m^2 i.v. over 2 hours and pemetrexed 500 mg/m^2 i.v. over 10 minutes on Day 1 of a 21day cycle. Cycles of treatment will be repeated every 3 weeks. Folic acid and B12 supplementation is obligatory.
  Interventions: Drug: Oxaliplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Oxaliplatin — Dose Regimen: 120 mg/m^2 on Days 1 every 21 days
  Other Names: Eloxatin™
Drug: Pemetrexed — Dose Regimen: 500 mg/m^2 on Days 1 every 21 days
  Other Names: Alimta™

SUMMARY:
The purpose of this study is:

* To find out if the chemotherapy treatment using Pemetrexed (Alimta) and Oxaliplatin (Eloxatin) given together will kill the cancer cells in the patient's body and shrink the size of their tumor. This may allow patients to live longer or decrease the frequency and/or severity of the symptoms caused by the cancer. Pemetrexed has been approved by the Food and Drug Administration (FDA) to treat Lung Cancer. Oxaliplatin has been approved by the FDA for the treatment of Colon Cancer. The combination of these two drugs has been used to treat patients with Non-Small Cell Lung Cancer in Italy but not yet in the USA

Other purposes of this study are:

* To better detail the toxic effects of this chemotherapy combination.
* To determine whether the level of specific gene and/or gene products (genes are genetic material that allows cells to make proteins such as enzymes) are useful to predict if this chemotherapy combination will work or not.

DETAILED DESCRIPTION:
Treatment Plan:

This is a non-randomized, two stage design, open-label Phase II trial in newly diagnosed patients with advanced or metastatic NSCLC who have previously received and failed adjuvant platinum-based chemotherapy for early stage, resected NSCLC.

Correlative Studies; Molecular correlative studies (genomic and proteomic) are included in this protocol. Prior to chemotherapy, all patients will undergo a biopsy of the safest and/or most accessible site of tumor in order to obtain tissue for mRNA measurements. Additionally, patients will undergo blood sampling prior to the start of chemotherapy and after 2 and 4 cycles of therapy in order to obtain plasma for the mass spectrometry analysis.

Patients, whose second and/or third specimen cannot be collected for any reason, will remain in the trial, and treatment will continue as outlined in the protocol.

Expected Number of Patients:

The number of patients was calculated according to the procedure described in the Sample Size Calculation section of the protocol. It is estimated that up to 50 patients will be enrolled to obtain the 43 evaluable patients needed to meet the statistical design of the study.

Method of Treatment Allocation:

A patient number will be assigned sequentially to each patient upon registration. The patient number and the patient initials are to be entered on each page of the Case Report Form.

Duration of Study for Each Patient:

All patients will be treated with up to 6 cycles of chemotherapy. However, at the discretion of the treating physician and principle investigator, patients may continue chemotherapy, beyond 6 cycles, until disease progression, intolerable toxicity, or the development of any study removal criteria. Patients will undergo an evaluation for extent of disease after every other treatment cycle.

Patients will be considered to be on-study for the duration of their treatment and during the 30 days following treatment discontinuation. Treatment discontinuation is defined as the last day of study treatment. All included patients will be followed up until recovery or stabilization of all adverse events or return to baseline condition. Patients who discontinue from the trial prior to experiencing disease progression will be followed monthly until demonstration of progressive disease.

Study Centers:

The H. Lee Moffitt Cancer Center will conduct this trial through the Moffitt Clinical Research Affiliate Network. Patients will be evaluated and the biopsy will be performed at the H. Lee Moffitt Cancer Center. Since all the chemotherapeutic drugs used in the protocol are FDA approved, and phase I and II safety data regarding this regimen has been published30,31, the chemotherapy may be administered at the patients' primary (referring) oncologists' office. Documentation of the administration of the chemotherapy will be obtained for record keeping purposes.

ELIGIBILITY:
Inclusion Criteria:

* History of completely resected NSCLC and adjuvant/neoadjuvant chemotherapy with platinum-based regimen
* Histologically/cytologically confirmed recurrence of NSCLC after curative therapy with surgery and adjuvant/neoadjuvant chemotherapy
* Must have measurable disease according to RECIST criteria
* ECOG Performance Score of 0-2 determined within 2 weeks prior to enrollment
* Expected survival > 12 weeks
* Adequate bone marrow function,as evidenced by:

  1. Absolute neutrophil count (ANC) > 1,500/µL
  2. Platelet count > 100,000/µL
  3. Hemoglobin > 8 g/dL (determined within 2 weeks prior to enrollment)
* Adequate renal function evidenced by:

  1. serum creatinine < 1.5 mg/dL OR
  2. calculated creatinine clearance >45 mL/min.
* Adequate hepatic function evidenced by:

  1. Serum total bilirubin < 1.5 mg/dL OR less than the upper limit of normal (ULN)
  2. Alkaline phosphatase < 3X the ULN for the reference lab (< 5X the ULN for patients with known hepatic or bony metastases)
  3. SGOT/SGPT < 3X the ULN for the reference lab (< 5X the ULN for patients with known hepatic metastases)
* Must be recovered from both acute and late effects of any prior surgery, radiotherapy, other antineoplastic therapy
* Signed informed written consent
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following last dose of study medication

Exclusion Criteria:

* Patients amenable to a "curative intent" therapeutic approach (re-resection with or without preoperative or postoperative therapy or chemoradiotherapy without surgery are not eligible for this study).
* An active infection or with fever > 101.00 F within 3 days of first scheduled day of protocol treatment
* Active CNS metastases. Patients with stable CNS disease, who have undergone radiotherapy (or surgery ± radiotherapy) at least 4 weeks prior to planned first protocol treatment and who have been on stable or decreasing dose of corticosteroids for >2 weeks are eligible
* Prior malignancy within the past 5 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with most recent evaluation no more than 4 weeks prior to entry.
* Any diagnosis of NSCLC occurring after 5 years of curative therapy (surgery plus adjuvant chemotherapy) for original NSCLC will be considered a second primary rather than a recurrence and will render patient ineligible for this study. An exception will be if both tumors are considered the same after a direct pathologic comparison if both, sponsor and investigator agree.
* Patients that at discretion of the PI have a second primary rather than metastasis are not eligible
* Known hypersensitivity to any of the components of oxaliplatin or pemetrexed.
* Patients receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment
* Patients who received radiotherapy to more than 33% of their bone marrow or received any radiotherapy within 4 weeks of entry
* Peripheral neuropathy ≥ Grade 2
* Patients pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed likely to interfere with patient's ability to sign informed consent, cooperate and participate in the study, or interfere with interpretation of the results.
* History of allogeneic transplant
* Known history of HIV or Hepatitis B or C infection. Patients with Hepatitis B carrier status only are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Chiappori, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: Single arm, two stage design Phase II study offered through the Moffitt Clinical Research Affiliate Network
Period: Overall Study
Arm/Group | Chemotherapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — study closed before treatment started | 1

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Responded to Treatment
Description: We planned to determine the Overall Response Rate (ORR = CR+PR) of this regimen according to RECIST Criteria.
Time Frame: Patient will continue study treatment until death, disease progression, unacceptable toxicity, patient refusal, or treatment delay > 3 weeks.
Population: Study closed before treatment started.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Time to Progression (TTP)
Description: We planned to calculate the median Time to Progression of all participants.
Time Frame: as for outcome 1
Population: Study closed before treatment started.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Who Experienced Toxicities
Description: We planned to determine the safety of the regimen (Drug Toxicities) assessed by NCI Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0)
Time Frame: as for outcome 1
Population: Study closed before treatment started.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Terminated due to slow accrual. Study closed before treatment started.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No